CLINICAL TRIAL: NCT01557634
Title: An Open-label, Single-centre, Randomised, 2-period Cross-over Study to Assess the Efficacy and Safety of Overnight Closed-loop Insulin Delivery Using Diluted Insulin in Comparison With Closed-loop With Non-diluted Insulin in Children With Type 1 Diabetes Aged 2 to 6 Years
Brief Title: Closing the Loop in Young Children With Type 1 Diabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daniela Elleri (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Daniela Elleri, Clinical Research Fellow, University of Cambridge
Organization: University of Cambridge (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: APCam10
Record Dates: First submitted 2012-03-14; First posted 2012-03-19 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2012-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed-loop with diluted insulin (Experimental): Insulin pump therapy using diluted insulin (20 IU/ml) will be driven by computer-based algorithm from 1700 on Day 1 until 0800 on Day 2
  Interventions: Procedure: Overnight closed-loop insulin delivery
- Closed-loop with non-diluted insulin (Active Comparator): Insulin pump therapy using standard non-diluted insulin (100 IU/ml) will be driven by computer-based algorithm from 1700 on Day 1 until 0800 on Day 2
  Interventions: Procedure: Overnight closed-loop insulin delivery

INTERVENTIONS:
Procedure: Overnight closed-loop insulin delivery — Basal insulin infusion rates on insulin pump will be directed by MPC algorithm using diluted versus non-diluted insulin

SUMMARY:
The incidence of type 1 diabetes (T1D) is increasing worldwide with evidence of most rapid increase in preschool children. Intensive control of blood glucose levels, although essential to protect against onset and progression of diabetes-related complications, faces unique challenges in toddlers and preschool children. A closed-loop system can enhance accuracy of insulin delivery and help people with T1D attain a tight glucose control avoiding the risk of hypoglycaemia. The main components of the system are a continuous glucose monitor (CGM), an insulin pump and a computer-based 'model predictive algorithm', which calculates the amount of insulin to be given by the insulin pump according to the CGM values. In the studies performed thus far the efficacy and safety of closed-loop glucose control were evaluated in children and adolescents aged 6 to 18 years. The results showed that closed-loop improved control of blood glucose and prevented nocturnal hypoglycaemia, as compared to the conventional insulin pump therapy. The objective of the current study is to extend the evaluation of closed-loop further to younger children aged 2 to 6 years, who may gain a great benefit from this novel therapy. The present study adopts an open-label, randomised, 2 period cross-over design whereby closed-loop insulin therapy using diluted insulin (20IU/ml)will be compared with closed-loop with standard insulin (100IU/ml)in 12 young children with T1D. Participants aged 2 to 6 years will be randomised for two overnight studies in a clinical research facility, during which glucose levels will be controlled by either the computer-based closed-loop algorithm using diluted insulin or by closed-loop with standard insulin. On both occasions, participants will receive a self-selected evening meal and closed-loop will run from 17:00 until 08:00am the following day. The study will take place at the Wellcome Trust Clinical Research Facility, Cambridge with participants recruited from paediatric diabetes clinics in England.

ELIGIBILITY:
Inclusion Criteria:

* The subject is between 2 and 6 years of age (inclusive)
* The subject has had type 1 diabetes, as defined by WHO criteria for at least 6 months
* The subject will be an insulin pump user and carers will have a good knowledge of insulin dose adjustment
* HbA1c below 12 % (108mmol/mol)

Exclusion Criteria:

* Non-type 1 diabetes mellitus including those secondary to chronic disease
* Any other physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results
* Current treatment with drugs known to interfere with glucose metabolism such as systemic corticosteroids
* Known or suspected allergy against insulin

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Time in target | Between 21:00 on Day 1 and 8:00 on Day 2
  Time spent with plasma glucose concentration in the target range (3.9-8.0mmol/L)

SECONDARY OUTCOMES:
Time below target | Between 21:00 on Day 1 and 8:00 on Day 2
  • Time spent with plasma glucose concentration below the target range (<3.9mmol/L)
Glucose variability | Between 21:00 on Day 1 and 08:00 on Day 2
  • Glucose variability as measured by standard deviation of glucose

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, Principal Investigator — University of Cambrigde
Locations (1):
- Wellcome Trust Clinical Research Facility, Addenbrooke's hospital, Cambridge, United Kingdom

REFERENCES:
- [Background] Hovorka R, Allen JM, Elleri D, Chassin LJ, Harris J, Xing D, Kollman C, Hovorka T, Larsen AM, Nodale M, De Palma A, Wilinska ME, Acerini CL, Dunger DB. Manual closed-loop insulin delivery in children and adolescents with type 1 diabetes: a phase 2 randomised crossover trial. Lancet. 2010 Feb 27;375(9716):743-51. doi: 10.1016/S0140-6736(09)61998-X. Epub 2010 Feb 4. PMID 20138357
- [Derived] Ruan Y, Elleri D, Allen JM, Tauschmann M, Wilinska ME, Dunger DB, Hovorka R. Pharmacokinetics of diluted (U20) insulin aspart compared with standard (U100) in children aged 3-6 years with type 1 diabetes during closed-loop insulin delivery: a randomised clinical trial. Diabetologia. 2015 Apr;58(4):687-90. doi: 10.1007/s00125-014-3483-6. Epub 2014 Dec 24. PMID 25537835
- [Derived] Elleri D, Allen JM, Tauschmann M, El-Khairi R, Benitez-Aguirre P, Acerini CL, Dunger DB, Hovorka R. Feasibility of overnight closed-loop therapy in young children with type 1 diabetes aged 3-6 years: comparison between diluted and standard insulin strength. BMJ Open Diabetes Res Care. 2014 Dec 11;2(1):e000040. doi: 10.1136/bmjdrc-2014-000040. eCollection 2014. PMID 25512874